CLINICAL TRIAL: NCT04030663
Title: The Effect of Periradial Injection of Papaverine Versus Nitroglycerine on Radial Artery Diameter Prior to Cannulation.
Brief Title: The Effect of Periradial Injection of Papaverine Versus Nitroglycerine on Radial Artery Diameter
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, ahmed said, lecture of anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FWA00015574
Record Dates: First submitted 2019-07-21; First posted 2019-07-24 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Radial Artery Injury Prevetion
MeSH Terms: interventions — Papaverine; Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- papaverine (Active Comparator)
  Interventions: Drug: papaverine
- nitroglycerine (Active Comparator)
  Interventions: Drug: nitroglycerine
- xlyocaine (Placebo Comparator)
  Interventions: Drug: xlyocaine

INTERVENTIONS:
Drug: papaverine — periradial injection of one of three drugs prior to cannulation of radial artery by 20 minutes and mesure the diamter of it by ultrasound
  Arms: papaverine
Drug: nitroglycerine — periradial injection of one of three drugs prior to cannulation of radial artery by 20 minutes and mesure the diamter of it by ultrasound
  Arms: nitroglycerine
Drug: xlyocaine — periradial injection of one of three drugs prior to cannulation of radial artery by 20 minutes and mesure the diamter of it by ultrasound
  Arms: xlyocaine

SUMMARY:
Compare the effect of periradial injection of papaverine versus nitroglycerine on radial artery diamter before cannulation of it in cardiac surgery.

DETAILED DESCRIPTION:
we want in this study to facilitate radial artery canulation and decrease the number of attemps of puncture which may lead to disappearance of the pulse.

The aim of this study is to compare the effect of adding papaverine to local anesthetic xylocaine versus adding nitroglycerine to it on the diameter and palpability of radial artery and if perioperative spasm will decrease significantly with one of these methods.

ELIGIBILITY:
Inclusion Criteria:

- Patients who will be included in the study are those scheduled for elective cardiac surgery who are hemodynamically stable.

Exclusion Criteria:

* Any patient with negative modified Allen test, atrioventricular block, glaucoma, altered liver function, unstable hemodynamics, emergency surgeries, and peripheral vascular disease.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
diameter of radial artery | 20 minutes
  after periradial injection of one of the drugs we will feel the radial artery pulse and record if there is a change in the palpatory score and mesure the diameter of the radial artery by ultrasound in cardiac surgery patients

SECONDARY OUTCOMES:
spasm of radial artery | 24 hours
  detect if there is postoperative spasm of radial artery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo, Benisuef, Egypt

IPD SHARING:
Plan to Share IPD: No